CLINICAL TRIAL: NCT02188134
Title: Quantifying the Attentive Behaviors of Older Adults During Over-the-counter Drug Selection
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Collaborators: Consumer Healthcare Products Association (Other)
Responsible Party: Principal Investigator, Laura Bix, Associate Professor, Michigan State University
Other Study IDs: MSU14-679
Record Dates: First submitted 2014-07-08; First posted 2014-07-11 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Older Adults (65 Years and Older)
Keywords: Adverse events,; adverse drug reactions,; medication error,; noncompliance
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Patient Compliance

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 65 and older: No intervention will be administered

SUMMARY:
Per-capita consumption of medication is higher in older adults than any other sector of the population. In fact, it has been estimated that although older adults comprise 13% of the population they take 34% of all prescriptions and 30% of the over-the-counter (OTCs) consumed in the US (National Council on Patient Information and Education, 2010). Given current trends in aging, the savings, freedom and flexibility that self-medicating provides, as well as the trends to switch prescription products to an OTC status, it is likely that older adults will increasingly turn to OTCs as part of their medical regimens for years to come (Hanlon, J et al, 2001).

In addition to the advantages that self-medicating offers, there are risks. These risks are more pronounced in older consumers, who are likely experiencing physiological changes (e.g. pharmacokinetics, pharmacodynamics, perceptual, cognitive and motor); this combines with a propensity for poly-pharmacy that escalates the likelihood of adverse drug reactions. It has also been suggested that low health literacy rates in older consumers detrimentally impact health and health outcomes in this population (Kutner et al., 2005 and Federman et al., 2009).

Despite the risks associated with improper OTC use, the critical importance of OTC labeling information (there is no learned intermediary), and the fact that older consumers are significantly more likely to experience an adverse drug reaction than younger adults, surprisingly little information exists about the decision making process older adults employ when selecting and using an OTC product.

We propose to recruit people 65 and older for an eye tracking study of mock OTC brands. The study has the following objectives:

1. To begin to garner insights regarding the proportion of subjects who closely examine (e.g. turn to the Drug Facts Label) the labeling of an OTC when deciding whether (or not) a drug is appropriate for them (based on their health history and current medications).
2. To quantify and compare the attentive behaviors to specific information (Specifically: name, active ingredient, symptom relief).
3. To quantify and compare the attentive behaviors to different formats of information (prominently featured information vs less prominently featured information).
4. To begin to benchmark whether or not older consumers make appropriate choices based on their current conditions and medication history.

DETAILED DESCRIPTION:
Eligibility Criteria 65 or older Administer own medications Legally sighted Purchase over-the-counter medications on occasion Be willing to share complete health history and complete list of all OTC and prescription medications Have transportation to one of two test sites (MSU Campus or Lansing Ingham County Building)

ELIGIBILITY:
Inclusion Criteria:

* 65 or older legally sighted administer own medication purchase OTC have transportation to one of two test sites Be willing to share a complete health history and complete list of medications

Exclusion Criteria:

* Legally blind Does not use OTC medications Less than 65 Does not administer own medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 65 and older self administer medication Purchase OTCs
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time in zone | Measure taken in a single session with participant
  Eye tracking will be done while mock OTCs appear on a computer screen, and participants will be asked to make a binary choice (yes/no) regarding whether (or not) the drug is safe choice for them at present.
  Treatments will appear in random order . Subjects will be asked to answer the question, "Assuming you have this condition, is this product appropriate for you?" for each of the twenty-seven trials while we track the movement of the eye.
  Zones for the analysis of the data include product name, symptom relief and active ingredient. Time in zone is the amount of time a subject's eye spends on the targeted information.
Time to first hit | Measure taken in a single session with participant
  Eye tracking will be done while mock OTCs appear on a computer screen, and participants will be asked to make a binary choice (yes/no) regarding whether (or not) the drug is safe choice for them at present.
  Treatments will appear in random order . Subjects will be asked to answer the question, "Assuming you have this condition, is this product appropriate for you?" for each of the twenty-seven trials while we track the movement of the eye.
  Zones for the analysis of the data include product name, symptom relief and active ingredient. Time to first hit is the measure of time it takes for a subject to fixate information in the zones described above.
Number of visual hits | Measure taken in a single session with participant
  Eye tracking will be done while mock OTCs appear on a computer screen, and participants will be asked to make a binary choice (yes/no) regarding whether (or not) the drug is safe choice for them at present.
  Treatments will appear in random order . Subjects will be asked to answer the question, "Assuming you have this condition, is this product appropriate for you?" for each of the twenty-seven trials while we track the movement of the eye.
  Zones for the analysis of the data include product name, symptom relief and active ingredient. Number of visual hits is the number of times the eye returns to a given information zone
Appropriate product selection | Measure taken in a single session with participant
  Eye tracking will be done while mock OTCs appear on a computer screen, and participants will be asked to make a binary choice (yes/no) regarding whether (or not) the drug is safe choice for them at present.
  Treatments will appear in random order . Subjects will be asked to answer the question, "Assuming you have this condition, is this product appropriate for you?" for each of the twenty-seven trials while we track the movement of the eye.
  Based on the self-reported history that is provided during a guided interview, and the medications that they have brought with them, an assessment will be made regarding the "correctness" of their response to whether or not the drug is an appropriate choice for them

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bix, PhD, Principal Investigator — Michigan State Univeristy
Locations (1):
- Packaging Building, East Lansing, Michigan, United States